CLINICAL TRIAL: NCT04558203
Title: The Relationship Between COVID-19 and Autoimmune Diseases, Lessons From Practice
Status: Completed | Type: Observational
Sponsor: ClinAmygate (Other)
Responsible Party: Sponsor
Other Study IDs: PR0014
Record Dates: First submitted 2020-09-19; First posted 2020-09-22 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Autoimmune suspected cases: Cases suspected to have autoimmune diseases
- non - autoimmune suspected cases: non - autoimmune suspected cases

SUMMARY:
The study explore the relationship between COVID-19 and the induction of autoimmune diseases.

This study comprises both retrospective and prospective components. The retrospective arm (2016-2019) was conducted to establish baseline incidence rates of autoimmune diseases (AIDs) prior to the COVID-19 pandemic. The prospective arm (2020-2024) involves the identification and longitudinal follow-up of newly diagnosed AID cases to evaluate disease progression, therapeutic response, and recurrence. Based on these data, the study will yield four distinct analyses:

1. trends in AID incidence before and after the COVID-19 pandemic,
2. the demographic and clinical profile of AID patients in the post-COVID-19 era,
3. the association between COVID-19 vaccine status and the development of AIDs, and
4. the clinical course, response to therapy, and long-term outcomes of AIDs in post-COVID patients compared to pre-pandemic cases.

DETAILED DESCRIPTION:
It has been suggested that the shared pathogenetic mechanisms and clinical-radiological aspects between the hyper-inflammatory diseases and Covid-19 may suggest that SARS-CoV-2 could act as a triggering factor for the development of a rapid autoimmune and/or autoinflammatory dysregulation, leading to the severe interstitial pneumonia, in genetic predisposed individuals.

The study is designed to investigate four primary objectives:

1. the incidence and trends of autoimmune diseases (AIDs) before and after the COVID-19 pandemic,
2. the association between COVID-19 vaccine status and the development of AIDs,
3. the clinical progression, treatment response, and recurrence of AIDs in post-COVID patients, and
4. the demographic and clinical profile, contributing factors, and spectrum of AID types identified during the post-pandemic period.

Retrospective data from 2016 to 2019 will be analyzed to establish baseline incidence rates, while prospective data from 2020 to 2024 will focus on new cases, vaccine exposure, clinical course, and patient characteristics.

The investigators hypothesize that:

1. the incidence of AIDs has increased in the post-COVID-19 era compared to the pre-pandemic period,
2. there is a positive association between COVID-19 vaccination and the onset of AIDs,
3. the clinical course and therapeutic response of AIDs in post-COVID patients differ from historical cases, and
4. unique demographic and clinical patterns characterize AID cases arising during the post-COVID period.

Accordingly, the study will yield four distinct analyses, each to be reported in a separate manuscript corresponding to the above objectives.

ELIGIBILITY:
Inclusion Criteria:

* all gender
* all age

Exclusion Criteria:

* Those who refused to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study population are all patients came to the center with or without symptoms and signs suspected to be AID during the study period
Sampling Method: Non-Probability Sample
Enrollment: 10510 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-01-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Incidence Rate of Autoimmune Diseasee | 2016-2024
  The number of new AID cases per 100,000 population before and after COVID-19, analyzed using retrospective and prospective data.
Disease severity | one week
  Severity as mild, moderate, severe according to type of AIDs
recurrence of AIDs | one year
  number of recurrence of the disease within the follow up period
response to therapy in the acute phase | within 4 weeks
  good response, weak response that need escalation of the dose of corticosteroids, no response

SECONDARY OUTCOMES:
recurrence as another auto-immune disease | Up to 4 years
  recurrence of different auto-immune disease
change in inflammatory markers | Two-months to Twelve months
  behavior of laboratory data of C-reactive protein, sedimentation rate, ferritine
incidence of other complications | Two-months to Twelve months
  incidence of other complications

CONTACTS AND LOCATIONS:
Overall Officials: Emad R Issak, MD, Principal Investigator — Asalam Center
Locations (1):
- Asalam, Maadi, Cairo Governorate, Egypt

REFERENCES:
- [Background] Ehrenfeld M, Tincani A, Andreoli L, Cattalini M, Greenbaum A, Kanduc D, Alijotas-Reig J, Zinserling V, Semenova N, Amital H, Shoenfeld Y. Covid-19 and autoimmunity. Autoimmun Rev. 2020 Aug;19(8):102597. doi: 10.1016/j.autrev.2020.102597. Epub 2020 Jun 11. No abstract available. PMID 32535093